CLINICAL TRIAL: NCT06094868
Title: A Single-arm, Open-label, Multicenter Phase II Clinical Study of Fruquintinib Combined With Sintilimab and XELOX in the First-line Treatment of Advanced Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Clinical Study of Fruquintinib Combined With Sintilimab and XELOX Regimen in the Treatment of Advanced Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Hua Wang, Director, Second Affiliated Hospital of Nanchang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-E1-GC002
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — HMPL-013; sintilimab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib in combination with Sintilimab and XELOX (Experimental): Fruquintinib: 4mg, QD, PO, D1-D14, Q3W; Sintilimab: weight < 60kg, 3mg/kg; weight≥60kg, 200 mg; I.V.， D1，Q3W； XELOX regimen: oxaliplatin: 130 mg/m2, ivgtt, D1, Q3W; Capecitabine: 1000 mg/m2, bid, D1-D14, Q3W; After 6 cycles of treatment, chemotherapy was given and maintenance treatment was given with fuquitinib combined with sindillizumab. The above medication regimen can be adjusted according to the adverse reaction tolerance of the subjects.
  * Maintenance of treatment until disease progression, or intolerable toxic reactions, or other conditions determined by the investigator
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib: 4mg, QD, PO, D1-D14, Q3W; Sintilimab: weight < 60kg, 3mg/kg; weight≥60kg, 200 mg; I.V.， D1，Q3W；. XELOX regimen: Oxaliplatin: 130 mg/m2, ivgtt, D1, Q3W; Capecitabine: 1000 mg/m2, bid, D1-D14, Q3W; After 6 cycles of treatment, chemotherapy was given and maintenance treatment was given with Fruquintinib combined with Sintilimab. The above medication regimen can be adjusted according to the adverse reaction tolerance of the subjects.
  * Maintenance of treatment until disease progression, or intolerable toxic reactions, or other conditions determined by the investigator
  Other Names: Sintilimab; Oxaliplatin; Capecitabine

SUMMARY:
To explore the efficacy and safety of Fruquintinib combined with Sintilimab and XELOX in the first-line treatment of unresectable advanced metastatic gastric or gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
To explore the progression-free survival (PFS), objective response rate (ORR), disease control rate (DCR), overall survival (OS), and safety of Fruquintinib combined with Sintilimab and XELOX in the first-line treatment of unresectable advanced metastatic gastric or gastroesophageal junctional adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood the study and voluntarily signed the informed consent;
2. Histologically and/or cytologically confirmed unresectable advanced gastric or gastroesophageal junction adenocarcinoma;
3. Age 18-75 (including 18 and 75 years old);
4. ECOG physical condition 0-1 score;
5. Locally advanced unresectable or metastatic gastric/gastroesophageal junction adenocarcinoma that has not received systemic therapy before (Note: Time from the end of previous (new) adjuvant chemotherapy/adjuvant radiotherapy to disease recurrence > 6 months);
6. For local lesions (non-target lesions), the time from the end of palliative treatment to random enrollment was > 2 weeks;
7. At least one measurable or evaluable lesion according to RECIST v1.1 criteria;
8. Negative Her2;
9. Expected survival ≥3 months;
10. The functions of vital organs during the first 14 days of enrollment met the following requirements:

    * Absolute neutrophil count ≥1.5×109/L;
    * Platelet ≥80×109/L;
    * Hemoglobin ≥90g/L;
    * Total bilirubin < 1.5 ULN;
    * ALT and AST < 2.5 ULN (< 5 ULN in patients with liver metastasis);
    * Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (CCr)≥60ml/min;
    * endogenous creatinine clearance > 50ml/min;
11. Female subjects of childbearing age or male subjects whose sexual partner is a female of childbearing age should take effective contraceptive measures throughout the treatment period and 6 months after the treatment period;
12. Good compliance, cooperate with follow-up.

Exclusion Criteria:

1. Failure to comply with the study protocol or study procedure;
2. Previous treatment with vascular endothelial growth factor receptor (VEGFR) inhibitors or previous treatment with immune checkpoint inhibitors;
3. Have had other malignancies within the past 5 years, except basal cell or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix;
4. Known presence of symptomatic central nervous system metastasis and/or cancerous meningitis. Participants with previously treated BMS may participate in the trial if their condition is stable (no evidence of radiographic progression at least 4 weeks prior to initial administration of the trial treatment), repeated radiographic studies confirm no evidence of new BMS or enlargement of the original BMS, and no steroid therapy is required at least 14 days prior to initial administration of the trial treatment. This exception does not include cancerous meningitis, which should be excluded regardless of whether it is clinically stable;
5. Had autoimmune disease or history of autoimmune disease within 4 weeks before enrollment;
6. Previously received allogeneic bone marrow transplantation or organ transplantation;
7. Uncontrolled malignant ascites (defined as ascites that cannot be controlled by diuretics or puncture as determined by the researcher);
8. Severe cardiovascular disease, including unstable angina pectoris or myocardial infarction, occurs within 6 months before the start of study treatment;
9. Subjects who are allergic to the investigational drug or any of its adjuncts;
10. Participated in other domestic unapproved or unmarketed drug clinical trials and accepted the corresponding experimental drug treatment within 4 weeks before enrollment;
11. Had a major surgical procedure (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of study therapy or expected to require major surgery during study therapy.
12. International Standardized Ratio (INR) > 1.5 or partially activated prothrombin time (APTT) > 1.5×ULN;
13. The investigator identified clinically significant electrolyte abnormalities;
14. Hypertension that could not be controlled by drugs before enrollment was defined as: systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg;
15. Poorly controlled diabetes mellitus was present before enrollment (fasting glucose concentration ≥CTCAE level 2 after formal treatment);
16. Had any disease or condition prior to enrollment that affected drug absorption, or the patient could not take fuquintinib orally;
17. Gastrointestinal diseases such as active ulcer of stomach and duodenum, ulcerative colitis, or active bleeding of unresectosed tumors, or other conditions that may cause gastrointestinal bleeding or perforation as determined by researchers before enrollment;
18. Patients with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding within 3 months > 30 mL, hematemesis, stool, stool blood), hemoptysis (within 4 weeks > 5 mL of fresh blood) or had a thromboembolic event (including stroke events and/or transient ischemic attacks) within 12 months;
19. Hepatic encephalopathy, hepatorenal syndrome or Child-Pugh grade B or more severe cirrhosis;
20. A history of intestinal obstruction or the following diseases: inflammatory bowel disease or extensive enterectomy (partial resection of the colon or extensive resection of the small intestine with chronic diarrhea), Crohn's disease, ulcerative colitis;
21. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months prior to enrollment; New York Heart Association (NYHA) Grades for Congestive Heart Failure > Level 2; Ventricular arrhythmias requiring medical treatment; LVEF (Left ventricular Ejection Fraction) < 50%;
22. Active or uncontrolled severe infection (≥CTCAE v5.0 grade 2 infection);
23. Known human immunodeficiency virus (HIV) infection. Known history of clinically significant liver disease, including viral hepatitis [Known hepatitis B virus (HBV) carriers must rule out active HBV infection, i.e., positive HBV DNA (>1×104 copies /mL or > 2000 IU/ml); known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL)];
24. Unmitigated toxicity higher than CTCAE v5.0 grade 1 due to any previous anticancer therapy, excluding alopecia, lymphocytopenia, and oxaliplatin grade ≤2 neurotoxicity;
25. Women who are pregnant (positive pregnancy test before medication) or breastfeeding;
26. Received blood transfusion therapy, blood products and hematopoietic factors, such as albumin and granulocyte colony-stimulating factor (G-CSF), within 14 days before enrollment;
27. Urine routine indicated urinary protein ≥2+, and 24-hour urinary protein volume > 1.0g;
28. Complications require long-term treatment with immunosuppressants or systemic or local use of immunosuppressive corticosteroids (> 10mg/ day prednisone or other therapeutic hormone);
29. Any other medical condition, clinically significant metabolic abnormality, physical abnormality or laboratory abnormality, which, in the investigator's judgment, reasonably suspects that the patient has a medical condition or condition that is not suitable for the use of the investigational drug (such as having seizures and requiring treatment), or which would affect the interpretation of the study results or place the patient at high risk。

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  The time from enrollment to disease progression or death Outcome 1
  Title:
  Progression-free survival (PFS)
  Description:
  The time from enrollment to disease progression or death

SECONDARY OUTCOMES:
Objective response rate (ORR) | During treatment
  Proportion of patients with complete or partial response
Disease control rate (DCR) | During treatment
  Proportion of patients assessed as having a complete response, partial response, or stable disease
Overall survival (OS) | Through study completion, an average of 1 year
  Patients were enrolled until their death from any cause
Security | Through study completion, an average of 1 year
  Safety was evaluated by adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Wang Hua, Director, Principal Investigator — Second Affiliated Hospital of Nanchang University